CLINICAL TRIAL: NCT04029194
Title: The Causal Effects of Old Age Pensions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Bureau of Economic Research, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 223749
Record Dates: First submitted 2019-04-26; First posted 2019-07-23 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-05

CONDITIONS: Aging
MeSH Terms: interventions — Insemination, Artificial, Heterologous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Behavioral: Assistance with old age pension application
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Assistance with old age pension application — The intervention will offer elderly assistance in applying for the old age pension.
  Arms: Treatment

SUMMARY:
Old age pensions are a common feature of welfare policy worldwide. However, little is known about the effect of these pensions on the recipients and their families. In this study, the investigators will partner with the government of Tamil Nadu, India to study the effects of old age pensions. Households with a member who is likely to be eligible for the pension but not currently receiving it will be assigned to either a treatment or control condition. Those assigned to treatment will receive assistance in applying for the pension. Investigators will track outcomes of the elderly and their family members for several years following the intervention.

In addition to the impact of pensions on economic and health outcomes, the study will also explore how pension receipt affects the elderly's ability to cope with the impact of the COVID crisis.

ELIGIBILITY:
Inclusion Criteria:

* Does not receive money from government scheme
* Over age 55
* Household does not own a house, or owns a kutcha house
* No member of the household is a working age male
* Household does not own any agricultural land, or household owns agricultural land and does not receive any income from agricultural activities
* No member of the household owns a car

Exclusion Criteria:

-

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1459 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Food consumption | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention.
  Value of consumption of food per capita in rupees over the last month. Households will be asked to report consumption of different food items over the last month in rupees; this will be added and divided by the number of household members to arrive at per capita values.
Goods and services consumption | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention.
  Yearly consumption on other goods and services in rupees. Households will be asked to report consumption of different goods and services over the last year in rupees; this will be added and divided by the number of household members to arrive at per capita values.
Self-assessment of financial wellbeing | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention.
  Household self-classification of its financial situation on 1-10 scale, with 1 being lowest and 10 being highest.
Food security | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention
  Whether any household member cut meals because of insufficient resources in the past year (0/1 variable)
Food security of elderly | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention
  Whether an elderly person cut meals because of insufficient resources in the past year (0/1 variable)
Difficulty in performing daily activities | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention.
  Participants will be asked over the last 30 days: how much difficulty they had in sitting for long periods, standing up from sitting down, getting up from lying down, standing for long periods, extending arms above shoulder level, washing whole body, getting dressed, getting to and using the toilet, taking care of household responsibilities, moving inside the home, walking 100 meters, walking long distances (1km), climbing a flight of stairs, stooping or kneeling, picking up things with fingers, carrying things, eating, getting where they want to go, concentrating on something for 10 minutes, learning a new task, and joining community activities. The scale is from 1-5, with 1 being no difficulty, 2 mild, 3 moderate, 4 severe, and 5 cannot do. The response for each activity will be converted to a z-score (subtract mean and divide by the standard deviation) and z-scores will be averaged to generate a composite index.
Basic and acute health | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention.
  Participants will be asked to report severity of basic and acute health conditions over the last 30 days. Two outcomes: difficulty seeing and difficulty hearing someone are measured on a scale from 1-5, with 1 being no difficulty, 2 mild, 3 moderate, 4 severe, and 5 cannot do. Three outcomes: any problems with mouth or teeth in the last 12 months, discomfort urinating, and any falls or injuries in the last 12 months will be measured on a yes or no basis. The response for each activity will be converted to a z-score (subtract mean and divide by the standard deviation) and z-scores will be averaged to generate a composite index.
Chronic health | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention.
  Participants will answer yes/no questions on whether they have any of the following health conditions: arthritis/rheumatism, stroke, chronic heart disease, hypertension and hypotension, diabetes, cancer, chronic lung disease, cholesterol, psychiatric illnesses, neurological disorders, kidney disease, liver disease. The response for each activity will be converted to a z-score (subtract mean and divide by the standard deviation) and z-scores will be averaged to generate a composite index.
Nutrition | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention.
  Participants will be asked if they lost ~5kg without wanting to in the past 6 months (0/1 variable), gets enough food every day (0/1 variable), and number of meals per day. Each will be converted into a z-score and averaged.
Mental health | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention.
  The geriatric depression index short form is used. Participants are asked yes/no questions: if they are satisfied with their lives, have dropped activities and interests, feel their life is empty, often get bored, in good spirits most of the time, afraid that something bad is going to happen to them, feel happy most of the time, often feel hopeless, prefer to stay at home, rather than going out and doing new things, have problems with memory, think it is wonderful to be alive, feel worthless, feel full of energy, feel lonely. Responses will be averaged.
Cognition | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention.
  Cognition status, based on performance in cognition "quiz", i.e. Mini Mental State Examination (MMSE).
Healthcare utilization | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention.
  Participants will be asked if they fell ill in the last 30 days, and, if yes, whether they used healthcare to deal with the illness (0/1); They will also be asked how much money (in rs.) they spent on health expenditure over the last 30 days. This will be converted into an index by averaging z-scores.
Loneliness | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention. Assessed during 3 phone surveys in March-December 2020, to gauge response to covid crisis.
  UCLA Loneliness scale short-form
Short-term food security during COVID | Assessed during 3 phone surveys in March-December 2020, to gauge response to covid crisis.
  Whether cut meals in the last week (0/1), whether they lack resources to buy food in the following week (0/1), whether their family skipped meals (0/1), and whether there was a shortage of food in their household during the last week (0/1). Averaged into an Anderson index.
Short-term mental health and loneliness during COVID | Assessed during 3 phone surveys in March-December 2020, to gauge response to covid crisis.
  Whether they often felt lonely in the last week (0/1), were afraid bad things would happen to them (0/1), felt their situation was hopeless (0/1). Averaged into an Anderson index.
Short-term medical access during COVID | Assessed during 3 phone surveys in March-December 2020, to gauge response to covid crisis.
  Whether they needed to but could not see a doctor in the last month (0/1), needed but could not get medication in the last month (0/1). Averaged into an Anderson index.
Short-term financial support during COVID | Assessed during 3 phone surveys in March-December 2020, to gauge response to covid crisis.
  Whether they continued to receive financial support from their family (0/1), whether family continued contributing to household expenses (0/1). Averaged into an Anderson index.
Short-term social distancing during COVID | Assessed during 3 phone surveys in March-December 2020, to gauge response to covid crisis.
  Whether they continued to work during lockdown (0/1), whether they planned to resume work during lockdown (0/1), whether they had in-person visits (0/1). Averaged into an Anderson index.
COVID vaccination rate | Assessed once, in a phone survey between March - May 2021, 8-11 months after intervention start.
  Whether they got the COVID vaccine.
Share of participants with COVID vaccine access | Assessed once, in a phone survey between March - May 2021, 8-11 months after intervention start.
  Whether they had someone take them to receive the COVID vaccine.

SECONDARY OUTCOMES:
Survival of elderly person | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention.
  Whether still living at time of follow-up survey (0/1 variable)
Labor supply of household members | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention.
  Whether employed (0/1 variable)
Labor supply of household members | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention.
  Amount of time spent working (days/week, hours/day)
Labor supply of household members | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention.
  Amount of income earned in rupees
Household structure 1 | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention.
  Number of adults in the household
Household structure 2 | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention.
  Number of children in the household
Assets | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention.
  Index of household asset ownership: car, two wheeler, TV, phone, refrigerator, washing machine, computer, air conditioner, internet.
Debt: household | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention.
  Whether any member of household has outstanding debt or a loan (0/1 variable)
Debt: elderly | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention.
  Whether elderly person has outstanding loan (0/1 variable)
Remittances | Assessed at 1 year, 3 years, 5 years, and at 7 years after intervention.
  Net amount of money sent (i.e. amount sent less amount received) to relatives outside of household in Rs.

CONTACTS AND LOCATIONS:
Locations (1):
- JPAL SA at IFMR, Chennai, Tamil Nadu, India

IPD SHARING:
Plan to Share IPD: No